CLINICAL TRIAL: NCT00956358
Title: Study on Systemic and Airway Cytokines and Oxidative Stress in Patients Undergoing Haemopoietic Stem Cell Transplantation (HSCT)
Brief Title: Study on Systemic and Airway Biomarkers in Haemopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Chung-Man HO, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 09-107
Record Dates: First submitted 2009-08-09; First posted 2009-08-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hematological Diseases
Keywords: bronchiolitis obliterans syndrome
MeSH Terms: conditions — Hematologic Diseases; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, buffy coat, red blood cell and exhaled breath condensate samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pre-HSCT: Haematological conditions requiring haemopoietic stem cell transplantation
- Post-HSCT with BOS: Occurence of bronchiolitis obliterans syndrome after haemopoietic stem cell transplantation
- Control: Healthy HSCT donors

SUMMARY:
Haemopoietic stem cell transplantation (HSCT) has become a major life-saving treatment for many haematological conditions, mostly malignancies.

However, there are lots of potential complications that hinder the long-term success of HSCT, in which bronchiolitis obliterans syndrome (BOS) is one of such serious complications. Basically, BOS represents a form of graft-versus-host immunological damage of small airways (bronchioles), leading to progressive narrowing of small airways and thus obstructive lung function abnormalities. With progressive loss of lung function in BOS, patients after HSCT can be complicated by intractable respiratory failure that results in mortality. Up until now, there is still no reliable way to accurately predict or detect BOS early to allow pharmacological interventions.

Therefore there is intense interest in the search for biomarkers that can help to predict the occurrence of BOS after HSCT. Apart from biomarkers (e.g., cytokines) in blood, there has been recent development in the sampling of airway lining fluid by a non-invasive method, i.e., collection of exhaled breath condensate (EBC). In airway diseases such as asthma or chronic obstructive pulmonary disease, EBC has been found to have various cytokines which can serve as potential biomarkers of disease activity. Since BOS is largely a small airway disease, it becomes logical to investigate the profile of biomarkers in EBC as predictors for BOS after HSCT.

Therefore this study has been designed to look into the role of biomarkers in blood and EBC in early detection of BOS after HSCT.

DETAILED DESCRIPTION:
Haemopoietic stem cell transplantation (HSCT) has revolutionized the treatment of both haematological and perhaps some solid malignancies. However, despite recent technological advancements, HSCT is still associated with significant mortality and morbidities.

Apart from various infective complications in early stage post-HSCT, bronchiolitis obliterans syndrome (BOS) has been a well-known late complication that can result in high mortality. It has been mostly associated with those who develop chronic graft-versus-host disease after allogeneic HSCT. Clinically, the diagnosis of BOS is largely based on demonstration of obstructive lung function abnormalities and air-trapping in computed tomography scan of thorax. Pathologically, bronchiolitis obliterans is characterized by both inflammatory and fibrotic reactions in the small bronchioles leading to subsequent obliteration. Upon diagnosis of BOS post-HSCT, inhaled corticosteroid (with or without bronchodilators) is commonly prescribed as anti-inflammatory agent, though with undocumented clinical efficacy. Unfortunately, there is still a lack of reliable biomarkers that can predict or allow early detection of BOS, preferably in the early and potentially reversible stage of development of BOS.

Apart from measuring circulating biomarkers in blood, exhaled breath condensate (EBC) has recently emerged as a non-invasive sampling method for real-time analysis and evaluation of oxidative stress biomarkers in the lower respiratory tract airways, especially in various lung diseases including asthma, chronic obstructive pulmonary disease, and lung cancer. As bronchiolitis obliterans is predominantly a disease of the small bronchioles, it is highly likely to be associated with changes in various inflammatory and oxidative stress biomarkers in EBC. However, the role of measuring EBC biomarkers in predicting the occurrence of BOS after HSCT has not been studied. Therefore, the current study aims to evaluate the temporal changes of various oxidative stress biomarkers and cytokines in EBC and blood in patients with haematological conditions who undergo allogeneic HSCT, with regard to the subsequent development of BOS.

ELIGIBILITY:
Inclusion Criteria:

* Haematological conditions requiring HSCT (either autologous or allogeneic with sibling donor), post-HSCT BOS, or healthy HSCT donors
* Life expectancy > 12 weeks

Exclusion Criteria:

* Respiratory failure requiring use of supplemental oxygen therapy
* Known airway diseases including asthma, chronic obstructive pulmonary disease and bronchiectasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Haematological conditions requiring HSCT and healthy HSCT donors will be identified from Bone Marrow Transplatation (BMT) Unit and post-HSCT patients with BOS will be identified from Respiratory Medicine clinics at Queen Mary Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2009-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Lung function indices | Every 3 months until either 18 months post-HSCT or diagnosis of BOS

CONTACTS AND LOCATIONS:
Overall Officials: Chung-man James Ho, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong